CLINICAL TRIAL: NCT00845936
Title: Metformin for Weight Control in Adolescents Taking Atypical Antipsychotics- Double Blind Placebo Controlled Study
Brief Title: Metformin for Weight Control in Adolescents Taking Atypical Antipsychotics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BeerYaakov Mental Health Center (Other Government)
Responsible Party: Pazit Leibovich, MD, BeerYaakov Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Metformin-38CTIL
Record Dates: First submitted 2009-02-15; First posted 2009-02-18 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Drug Induced Weight Gain
Keywords: Atypical antipsychotics; Weight; adolecsents; pediatric; Metformin
MeSH Terms: conditions — Body Weight | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): 850 mg of Metformin bid
  Interventions: Drug: Metformin
- placebo (Placebo Comparator): Tablets Identical to Metformin, bid
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 850 mg bid

SUMMARY:
Atypical antipsychotics (AA) are broadly used to treat a variety of psychiatric and neurological disorders in children and adolescents. Weight gain is a common side effect of these drugs. AA induced weight gain can be the cause of the metabolic syndrome which is a major health concern, as well as cancer and significant psychological disorders. Weight gain may also lead to low compliance with AAs.

A number of studies have been conducted in order to find a way to prevent, reduce or reverse AA induced weight gain in children and adolescents, but so far there is no commonly accepted treatment for the problem.

Metformin is an antihyperglycemic drug, approved by the FDA for treatment of type 2 diabetes in children older than 10 years of age. The drug usually does not cause hypoglycemia, even in high dosage. Contraindications include renal impairment, hepatic disease, a past history of lactic acidosis (of any cause), cardiac failure requiring pharmacological therapy, or chronic hypoxic lung disease. The drug also should be discontinued temporarily prior to the administration of intravenous contrast media and prior to any surgical procedure. The reported incidence of lactic acidosis during metformin treatment is less than 0.1 cases per 1000 patient-years, and the mortality risk is even lower.

Acute side effects of metformin, which occur in up to 20% of patients, include diarrhea, abdominal discomfort, nausea, metallic taste, and anorexia. These usually can be minimized by increasing the dosage of the drug slowly, when indicated, and taking it with meals. Intestinal absorption of vitamin B 12 and folate often is decreased during chronic metformin therapy, and calcium supplements reverse the effect of metformin on vitamin B12 absorption.

Three studies have studied the effect of metformin on weight gain secondary to use of AAs in adults and 3 other studies studied the effect of metformin in children and adolescents. Most of these studies have proved the drug to be efficient. No serious side effects have been demonstrated in any of these studies.

Objective- To assess the effect of metformin on body weight of children and adolescents treated by AAs.

Setting- recruitment and follow up would take place in the pediatric ward and outpatient clinic at the Ness- Tziona Mental Health Center.

Participants- 30 adolescents aged 12- 20 years old, treated with AAs, who are overweight as defined by more than 10% of what is expected according to age and height.

Importance of the Study

1. Identify a medication capable of reducing or preventing weight gain by an AA agent.
2. Identify an agent capable of improving compliance due to lower side-effect profile of AAs.

ELIGIBILITY:
Inclusion Criteria:

* 12-20 year olds treated by atypical antipsychotics
* weight gain of more than 10% than expected for age
* Overweight of more than 10% than expected for age and height

Exclusion Criteria:

* Physical conditions requiring pharmacological treatment
* Changes in drug type or dosage 2 months before the trial, except for 25% changes in dosage

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 12 weeks

SECONDARY OUTCOMES:
BMI, Weist circumstance, Blood pressure,Blood cholesterol,Fasting blood glucose and Insulin, Leptin levels. For safety- B12, Folate, lactate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beer-Yaacov MHC, Beer Yaacov, Israel